CLINICAL TRIAL: NCT01362647
Title: A Non-interventional / Observational Study on Postoperative Residual Curarisation at Arrival in the Post-anesthesia Care Unit After Spontaneous Recovery or After Reversal of the Neuromuscular Block
Brief Title: Postoperative Residual Curarisation at Arrival in the Post-anesthesia Care Unit
Status: Completed | Type: Observational
Sponsor: Onze Lieve Vrouw Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Guy Cammu, MD, PhD, OLV Hospital, Aalst, Belgium
Other Study IDs: B126201110617; IISP ID 39443 (Other Grant/Funding Number: MSD (Merck Sharp & Dohme))
Record Dates: First submitted 2011-05-25; First posted 2011-05-30 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2011-10

CONDITIONS: Postoperative Residual Curarisation; Postoperative Hypoxemia; Postoperative Airway Obstruction
Keywords: Muscle Relaxation
MeSH Terms: conditions — Delayed Emergence from Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: neuromuscular transmission monitoring — The acceleromyographic responses of the adductor pollicis muscle as percent of the train-of-four (TOF%) on stimulation of the ulnar nerve by means of TOF-Watch®, Organon Ireland Ltd., a division of MSD, Swords, Co., Dublin, Ireland.
Procedure: Pulse oximetry measurement — Pulse oximetry will be measured continuously throughout the PACU admission, and SpO2 values will be recorded at 1-min intervals for the first 30 min.

SUMMARY:
Several studies have documented that neuromuscular block often persists in the postanesthesia care unit (PACU). Residual paralysis is associated with postoperative complications such as hypoxia, weakness, and respiratory failure. The data in the current literature on residual paralysis in the PACU were almost exclusively obtained with acetylcholinesterase inhibitors as they were the only reversal agents available prior to the introduction in clinical practice of sugammadex (Bridion®) in the European Union and in some other countries, except for the USA. Reassessment of practice in this regard is relevant, now that sugammadex (Bridion®) has become available in our country since 2009.

This study is an observational/non-interventional, non-randomized study involving adult patients undergoing different types of elective surgical procedures requiring general anesthesia with neuromuscular blocking drugs (NMBDs). Administration of NMBDs and reversal agents (as well as all drugs which will be used during anesthesia) will be performed in accordance with routine anesthetic practice.

The study population will comprise about 600 surgical patients. Immediately after the patients' arrival in the PACU, a study nurse will record the acceleromyographic responses of their adductor pollicis muscle as percent of the train-of-four (TOF%) on stimulation of the ulnar nerve. A TOF of 90% will be used as cut-off value to exclude residual paralysis. Pulse oximetry (SpO2) will be measured continuously throughout the PACU admission, and SpO2 values will be recorded at 1-min intervals for the first 30 min. PACU nurses caring for the patient will document the occurrence of any of the following events during the first 30 min of PACU admission: the number of episodes of hypoxemia (SpO2<90%), the lowest SpO2 observed by nursing staff, the requirement for either tactile or verbal stimulation to maintain SpO2 greater than 90%, and any clinical evidence of airway obstruction.

The primary objective is to evaluate the incidence of postoperative residual curarisation at PACU arrival in patients reversed with sugammadex (Bridion®), neostigmine and in case of spontaneous recovery.

The secondary objectives are to evaluate:

* Oxygen saturation (SpO2) at PACU arrival
* Possible episodes of SpO2 <90% in the PACU
* Airway maneuvers and/or stimulation required to maintain SpO2 >90% in the PACU
* Need for re-intubation.

DETAILED DESCRIPTION:
• Background & Rationale: Several studies have documented that neuromuscular block often persists in the PACU, even with the administration of acetylcholinesterase inhibitors. Postoperative residual curarisation ranges between 4 and 50% depending on the diagnostic criteria, the type of non-depolarizing neuromuscular blocking drug (NMBD), the administration of a reversal agent, and the use of neuromuscular monitoring. Residual paralysis is associated with postoperative complications such as hypoxia, weakness, and respiratory failure. However, these complications may have many other causes so that the role of neuromuscular block is often unrecognized. Thus, it is important to manage neuromuscular block and have a strategy to prevent, diagnose, and treat residual paralysis, with neuromuscular monitoring and reversal of neuromuscular block in routine anesthetic practice. The data in the current literature on residual paralysis in the PACU were almost exclusively obtained with acetylcholinesterase inhibitors as they were the only reversal agents available prior to the introduction in clinical practice of sugammadex (Bridion®) in the European Union and in some other countries, except for the USA. Reassessment of practice in this regard is relevant, now that sugammadex (Bridion®) has become available in our country since 2009.

Five years ago a similar exploratory, non-interventional, non-randomized study took place in Belgium. This previous study will help to assess the two different periods (2005-2011) in terms of management of neuromuscular block in the operating room of a large regional community hospital.

• Study Design: This is an observational/non-interventional, non-randomized study involving adult patients undergoing different types of elective surgical procedures requiring general anesthesia with NMBDs. This study will reflect real life clinical practice. The anesthetic technique in terms of drugs and type of monitoring used will be the entire responsibility of the anesthesiologist.

All study activities will be consistent with EU directive 2001/20/EC for non-interventional studies (also known as observational/non-interventional studies).

Administration of NMBDs and reversal agents (as well as all drugs which will be used during anesthesia) will be performed in accordance with routine anesthetic practice; will follow good clinical practice and labeling of drugs. No other interventional means, methods or procedures are scheduled than those for routine care of the patient. Furthermore, there will be no additional visits to the hospital or a mandatory visit schedule, deviating from normal clinical practice.

• Study Flowchart: On arrival to the PACU, 3 l/min oxygen will be applied to all subjects by a nasal cannula. Baseline oxygen saturation values are recorded 1 min after application of the oxygen. Immediately after the patients' arrival in the PACU, a study nurse will record their tympanic temperatures and the acceleromyographic responses of their adductor pollicis muscle as percent of the train-of-four (TOF%) on stimulation of the ulnar nerve (TOF-Watch®, Organon Ireland Ltd., a division of MSD, Swords, Co., Dublin, Ireland). The stimulus current will be set in the range 25-35 mA for tolerance purpose without compromising the results. Two consecutive TOF measurements (separated by 15 s) will be obtained, and the average of the 2 values will be recorded. If measurements differ by >10%, additional TOF measurements will be obtained (up to 4 TOF values), and the closest 2 ratios averaged. A TOF of 90% will be used as cut-off value to exclude residual paralysis. Pulse oximetry will be measured continuously throughout the PACU admission, and SpO2 values will be recorded at 1-min intervals for the first 30 min. PACU nurses caring for the patient will document the occurrence of any of the following events during the first 30 min of PACU admission: the number of episodes of hypoxemia (SpO2<90%), the lowest SpO2 observed by nursing staff, the requirement for either tactile or verbal stimulation to maintain SpO2 greater than 90%, and any clinical evidence of airway obstruction. Patient demographic data, type of surgical procedure, duration of anesthesia, as well as data collected relating to neuromuscular management, will be recorded and stored on a PC.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* Informed consent signed;
* Admission for elective surgery;
* Administration of non-depolarizing NMBDs during surgery;
* Tracheal intubation

Exclusion Criteria:

* Evidence of renal, hepatic, metabolic, and/or neuromuscular disorders
* Ejection fraction <20%
* Admission for emergency surgery; or cardiothoracic surgery
* Reoperation during the same hospital admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will comprise about 600 surgical patients (the first 600 inpatients and outpatients scheduled for anesthesia during the study period who meet the study criteria).
Sampling Method: Non-Probability Sample
Enrollment: 625 (Actual)
Dates: Start 2011-05; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
incidence of postoperative residual curarisation | Immediately after the patients' arrival in the post-anesthesia care unit (<5 min after arrival), two consecutive neuromuscular transmission measurements (separated by 15 s) will be obtained, and the average of the 2 values will be recorded.
  incidence of postoperative residual curarisation (PORC) defined by a train-of-four (TOF) ratio < 0,9 at post-anesthesia care unit (PACU) arrival

SECONDARY OUTCOMES:
Possible episodes of SpO2 <90% in the PACU | During the first 30 min of PACU admission
Airway maneuvers and/or stimulation required to maintain SpO2 >90% in the PACU | During the first 30 min of PACU admission
  the requirement for either tactile or verbal stimulation to maintain SpO2 greater than 90%, and any clinical evidence of airway obstruction
Need for re-intubation | During the first 30 min of PACU admission

CONTACTS AND LOCATIONS:
Overall Officials: Guy Cammu, MD, PhD, Principal Investigator — OLV Hospital, Aalst, Belgium
Locations (1):
- OLV Hospital, Aalst, Belgium

REFERENCES:
- [Background] Cammu G, De Witte J, De Veylder J, Byttebier G, Vandeput D, Foubert L, Vandenbroucke G, Deloof T. Postoperative residual paralysis in outpatients versus inpatients. Anesth Analg. 2006 Feb;102(2):426-9. doi: 10.1213/01.ane.0000195543.61123.1f. PMID 16428537